CLINICAL TRIAL: NCT02054754
Title: Assessment of Safety, Tolerability and Pharmacokinetics of Single Doses of Oral Dexanabinol in Healthy Subjects
Brief Title: Assessment of Single Doses of Oral Dexanabinol in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: e-Therapeutics PLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ETS2101-101
Record Dates: First submitted 2013-11-20; First posted 2014-02-04 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Safety; Tolerability; Pharmacokinetics; Cancer
Keywords: Dexanabinol; Oral; Safety; Tolerability; Pharmacokinetics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Dexanabinol Dose Level 1 (Experimental): Single oral dose of dexanabinol
  Interventions: Drug: Dexanabinol Dose Level 1
- Dexanabinol Dose Level 2 (Experimental): Single oral dose of dexanabinol
  Interventions: Drug: Dexanabinol Dose Level 2
- Dexanabinol Dose Level 3 (Experimental): Single oral dose of dexanabinol
  Interventions: Drug: Dexanabinol Dose Level 3
- Dexanabinol Dose Level 4 (Experimental): Single oral dose of dexanabinol
  Interventions: Drug: Dexanabinol Dose Level 4
- Dexanabinol Dose Level 5 (Experimental): Single oral dose of dexanabinol
  Interventions: Drug: Dexanabinol Dose Level 5
- Placebo (Placebo Comparator): Single oral dose of matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexanabinol Dose Level 1 — Oral formulation of dexanabinol
  Other Names: ETS2101
  Arms: Dexanabinol Dose Level 1
Drug: Dexanabinol Dose Level 2 — Oral formulation of dexanabinol
  Other Names: ETS2101
  Arms: Dexanabinol Dose Level 2
Drug: Dexanabinol Dose Level 3 — Oral formulation of dexanabinol
  Other Names: ETS2101
  Arms: Dexanabinol Dose Level 3
Drug: Dexanabinol Dose Level 4 — Oral formulation of dexanabinol
  Other Names: ETS2101
  Arms: Dexanabinol Dose Level 4
Drug: Dexanabinol Dose Level 5 — Oral formulation of dexanabinol
  Other Names: ETS2101
  Arms: Dexanabinol Dose Level 5
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the safety and observe the pharmacokinetics (distribution and elimination of the drug) of the compound dexanabinol (ETS2101) in healthy male subjects following a single oral dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 18 to 45 years
* Body mass index 18.0 to 32.0 kg/m2, or if outside the range, considered not clinically significant by the investigator

Exclusion Criteria:

* Participation in a clinical research study within the previous 3 months
* Current smokers and those who have smoked within the last 12 months
* History of any drug or alcohol abuse in the past 2 years

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Evans, MD, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Nottingham, Nottinghamshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexanabinol Dose Level 1: Single oral dose of dexanabinol at Dose Level 1
  Dexanabinol: Oral formulation of dexanabinol
- Dexanabinol Dose Level 2: Single oral dose of dexanabinol at Dose level 2
  Dexanabinol: Oral formulation of dexanabinol
- Dexanabinol Dose Level 3: Single oral dose of dexanabinol at Dose level 3
  Dexanabinol: Oral formulation of dexanabinol
- Dexanabinol Dose Level 4: Single oral dose of dexanabinol at Dose level 4
  Dexanabinol: Oral formulation of dexanabinol
- Dexanabinol Dose Level 5: Single oral dose of dexanabinol at Dose level 5
  Dexanabinol: Oral formulation of dexanabinol
- Placebo: Single oral dose of matching placebo
  Placebo
Period: Overall Study
Arm/Group | Dexanabinol Dose Level 1 | Dexanabinol Dose Level 2 | Dexanabinol Dose Level 3 | Dexanabinol Dose Level 4 | Dexanabinol Dose Level 5 | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 10
Completed | 6 | 6 | 6 | 6 | 6 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy male subjects between 18 and 45 years of age with a body mass index between 18.0 and 32.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator.
Groups:
- Dexanabinol: Single oral dose of dexanabinol
  Dexanabinol: Oral formulation of dexanabinol
- Total: Total of all reporting groups
Arm/Group | Dexanabinol | Placebo | Total
Number analyzed (Participants) | 30 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (8.5) | 28.1 (8.3) | 31.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability Based on the Number of Participants With Adverse Events and Comparison of Baseline and Post Dose Parameters
Description: Safety and tolerability based on the number of participants with adverse events. Assessment and comparison to baseline of the following:
  * Physical exam
  * Safety bloods and urinalysis
  * 12-lead ECG
  * Vital signs
Time Frame: Participants will be followed until follow up visit, 6-11 days after dosing
Measure: Number; unit: participants
Arm/Group | Dexanabinol | Placebo
Number analyzed (Participants) | 30 | 10
participants | 9 | 1

2. Secondary Outcome: Area Under the Curve of the Compound Dexanabinol (ETS2101) From Pre-dose up to 48 Hours Post Dose
Description: Pharmacokinetic parameters will be assessed in a blinded fashion at the end of each cohort, prior to dose escalation.
Time Frame: Pre-dose, 0.5,1,1.5,2,3,4,5,6,8,10,12,16,24,36,48 hours post dose
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Dexanabinol Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 6
ng.h/mL | 37.5 (0) | 61.3 (75.7) | 109 (102.7) | 226 (50.7) | 192 (68.6)

3. Other Pre Specified Outcome: Pharmacodynamic Biomarker Assessment
Description: Blood samples taken and analysed for the purposes of the identification and quantification of pharmacodynamic biomarkers pre-dose and at several points after dosing.
Time Frame: Pre-dose, 1, 6 and 24 hours post dose
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Dexanabinol Dose Level 1; Dexanabinol Dose Level 2; Dexanabinol Dose Level 4; Dexanabinol Dose Level 5: Single oral dose of dexanabinol
  Dexanabinol: Oral formulation of dexanabinol
- Dexanabinol Dose Level 3: Single oral dose of dexanabinol
  Dexanabinol: Oral formuulation of dexanabinol
Arm/Group | Dexanabinol Dose Level 1 | Dexanabinol Dose Level 2 | Dexanabinol Dose Level 3 | Dexanabinol Dose Level 4 | Dexanabinol Dose Level 5 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 3/6 | 1/6 | 1/6 | 3/6 | 1/6 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexanabinol Dose Level 1 (N=6) | Dexanabinol Dose Level 2 (N=6) | Dexanabinol Dose Level 3 (N=6) | Dexanabinol Dose Level 4 (N=6) | Dexanabinol Dose Level 5 (N=6) | Placebo (N=10)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculo-skeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other